CLINICAL TRIAL: NCT07296445
Title: LATITUDE - A Phase 3, Randomized, Open-Label, 3-Cohort, 2-Period, 2-Sequence, Crossover Trial to Evaluate the Pharmacokinetics, Safety, and Efficacy of Oral Arsenic Trioxide Versus Intravenous Arsenic Trioxide for Consolidation Therapy in Participants With Newly Diagnosed, Non-High-Risk, Acute Promyelocytic Leukemia
Brief Title: A Trial to Investigate Whether Oral Arsenic Trioxide Is Similar to Intravenous Arsenic Trioxide in Pharmacokinetics, Safety, and Efficacy (LATITUDE/SDKARS-301)
Acronym: LATITUDE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SDK Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SDKARS-301; 2025-524329-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-16; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Acute Promyelocytic Leukemia (APL); Acute Promyelocytic Leukaemia; Acute Promyelocytic Leukemia With PML-RARA; Acute Promyelocytic Leukemia With t(15;17)(q24.1;q21.2); PML-RARA; APL; Acute Promyelocytic Leukemia; Leukaemia; Leukemia Acute Promyelocytic Leukemia (APL); Leukemia, Acute
Keywords: Oral Arsenic Trioxide; Oral ATO
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute; Leukemia | interventions — Arsenic Trioxide; Tretinoin

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, 3-Cohort, 2-Period, 2- Sequence, Crossover Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Cohort A (Experimental): Participants will receive Oral ATO 0.15 mg/kg daily × 5 days a week from Weeks 1 to 4 in the first three 8-week cycles, IV ATO 0.15 mg/kg daily (2-hour infusion) × 5 days in Week 1 of Cycle 4, and oral ATO 0.15 mg/kg daily × 5 days a week from Weeks 2 to 4 of Cycle 4. All adult participants will receive ATRA 45 mg/m2/day in 2 divided doses as background treatment 7 days a week for 2 weeks on and 2 weeks off (Weeks 1, 2, 5 and 6 of each 8-week cycle) beginning in Cycle 1 and ending after Cycle 4 Week 2
  Interventions: Drug: Oral ATO; Drug: IV Arsenic Trioxide; Drug: all-trans retinoic acid (ATRA)
- Part 1: Cohort B (Active Comparator): Participants will receive IV ATO 0.15 mg/kg daily (2-hour infusion) × 5 days a week from Weeks 1 to 4 in the first three 8-week cycles, oral ATO 0.15 mg/kg daily × 5 days in Week 1 of Cycle 4, and IV ATO 0.15 mg/kg daily (2-hour infusion) × 5 days a week from Weeks 2 to 4 of Cycle 4. All adult participants will receive ATRA 45 mg/m2/day in 2 divided doses as background treatment 7 days a week for 2 weeks on and 2 weeks off (Weeks 1, 2, 5 and 6 of each 8-week cycle) beginning in Cycle 1 and ending after Cycle 4 Week 2
  Interventions: Drug: Oral ATO; Drug: IV Arsenic Trioxide; Drug: all-trans retinoic acid (ATRA)
- Part 2: Cohort C (Experimental): Participants will receive Oral ATO 0.15 mg/kg daily × 5 days a week from Weeks 1 to 4 of four 8-week cycles. All adult participants will receive ATRA 45 mg/m2/day in 2 divided doses as background treatment 7 days a week for 2 weeks on and 2 weeks off (Weeks 1, 2, 5 and 6 of each 8-week cycle) beginning in Cycle 1 and ending after Cycle 4 Week 2
  Interventions: Drug: Oral ATO; Drug: all-trans retinoic acid (ATRA)

INTERVENTIONS:
Drug: Oral ATO — Oral Arsenic Trioxide
Drug: IV Arsenic Trioxide — Intravenous Arsenic Trioxide
  Arms: Part 1: Cohort A; Part 1: Cohort B
Drug: all-trans retinoic acid (ATRA) — all-trans retinoic acid (ATRA)

SUMMARY:
LATITUDE: A Phase 3, Randomized, Open-Label, 3-Cohort, 2-Period, 2- Sequence, Crossover Trial to Evaluate the Pharmacokinetics, Safety, and Efficacy of Oral Arsenic Trioxide Versus Intravenous Arsenic Trioxide for Consolidation Therapy in Participants With Newly Diagnosed, Non-High Risk, Acute Promyelocytic Leukemia

Rationale:

SDK Therapeutics is developing an oral formulation of arsenic trioxide (ATO) for the treatment of acute promyelocytic leukemia (APL). Patients with APL are usually treated with arsenic trioxide (ATO) through an IV along with all-trans retinoic acid (ATRA) taken by mouth. Receiving ATO through an IV requires patients with APL to go to the hospital a lot and get long treatments (sometimes every day over a year of treatment). This can be hard and uncomfortable. If ATO can be taken by mouth, it would be much easier for patients and their families.

Objective:

The main objective is to show that the body absorbs the same amount of ATO whether it's taken by mouth or through an IV. Other objectives include checking if ATO taken by mouth works just as well, causes fewer heart problems, is safe, and improves quality of life compared with ATO given through an IV.

Main trial endpoints:

The main endpoint being measured is how much ATO is in the blood after 5 doses. Another important endpoint is how many patients have no signs of cancer in their blood after 3 rounds of treatment.

Secondary trial endpoints:

Other things being measured include: whether patients stay cancer-free over 2 years; changes in heart rhythm; side effects and lab test results; how patients feel during treatment; how much of ATO is in the blood; and how often patients feel bothered by side effects.

Trial design:

This is an open-label study, meaning everyone knows which treatment they are getting. Patients will get 4 rounds of treatment, each lasting 8 weeks. After that, patients will have check-ups every 3 months to assess safety and disease status for a total of 2 years.

Trial population:

The study includes adults and teens (12 years and older) who have APL, are not high-risk, and have already finished the first part of their treatment (induction) with IV ATO and ATRA.

Interventions:

There are 3 groups in the study:

Cohort A: Takes 0.15 mg/kg Oral ATO for 3 rounds, then switches to 0.15 mg/kg IV ATO for part of the 4th round.

Cohort B: Takes 0.15 mg/kg IV ATO for 3 rounds, then switches to 0.15 mg/kg Oral ATO for part of the 4th round.

Cohort C: Takes 0.15 mg/kg Oral ATO for all 4 rounds.

All cohorts also take 45 mg/m2/day ATRA during certain weeks of each round. Doctors will assess efficacy by checking bone marrow samples before and during treatment to see if the cancer is gone. Special lab tests will be used to look for cancer cells. Safety will be assessed by checking for side effects using blood tests, heart tests, physical exams, and other health checks. Quality of life will be assessed by the patients who will fill out surveys about how they feel during treatment and how much the side effects bother them. The study will also look at how often patients need to go to the doctor or hospital; how treatment affects daily life and work; and how satisfied patients are with their treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have diagnosis of newly diagnosed non-high risk APL with a WBC count at diagnosis ≤ 10,000 cells/µL, completed induction with ATO/ATRA and achieved morphologic CR with hematologic recovery
* Eastern Cooperative Oncology Group performance status ≤2
* Adequate liver, kidney, and cardiac function
* Have a life expectancy of at least 9 months
* Negative serum pregnancy test

Key Exclusion Criteria:

* Diagnosis of relapsed or refractory APL.
* Fridericia's corrected QT interval (QTcF) >450 milliseconds (males) and >460 milliseconds (females)
* Any gastrointestinal (GI) issue likely to affect oral drug absorption/metabolism or inability to swallow oral medication
* Prior malignancy or currently receiving treatment for a non-APL malignancy, with the following exceptions: basal cell or squamous cell skin cancer treated with surgical resection, in situ cervical cancer, localized prostate cancer or breast cancer treated with hormone therapy or surgical resection, or other cancer from which the participant has been disease free for at least 2 years.
* Pregnant or nursing females or is of reproductive potential and unwilling to comply with contraceptive requirements.
* Participant has known active or chronic hepatitis B or active hepatitis C (HCV) infection or human immunodeficiency virus (HIV)-positive with detectable viral load.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic exposure (amount of ATO in the blood) | At the end of Cycle 4, Week 1 (Each cycle is 8 weeks)
  Total 5-dose plasma AsIII AUC

SECONDARY OUTCOMES:
Molecular Complete Response (molCR) rate | At the end of 3 Cycles of treatment (each cycle is 8 weeks)
  molCR rate, defined as negative/undetected for PML:RARα by RT-qPCR
Relapse-Free Survival (RFS) | Assessed for up to 2 years after the first dose of treatment, or until disease progression/relapse or death, whichever occurs first.
  2-year Relapse Free Survival (RFS)
Change in Fridericia-corrected QT interval (ΔQTcF interval) | At the end of Cycles 3 and 4 (each cycle is 8 weeks)
  Difference in QTcF between collected values
Adverse events | Up to 9 months
  Frequency, severity, and relatedness of adverse events.
Cardiac AEs related to elevated QTcF | Up to 9 months
  Number of prolonged QTcF interval or other arrhythmias per CTCAE
Pharmacokinetic profile | At the end of Cycle 4, week 1 (Each cycle is 8 weeks)
  Peak Plasma Concentration (Cmax)
Patient Reported Outcomes | Up to 9 months
  Change from baseline as measured by the EORTC QLQ-C30
Patient Reported Outcomes | Up to 9 months
  Proportion of time "bothered by side-effects" as measured by the FACT-GP5

IPD SHARING:
Plan to Share IPD: Undecided